CLINICAL TRIAL: NCT03472014
Title: A Special Access Program for the Prophylactic Vaccination With IMVAMUNE® for Personnel Working Directly With or in the Vicinity of Replicating Vaccinia Virus
Brief Title: Special Access Program IMVAMUNE®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: POX-MVA-03x
Record Dates: First submitted 2018-03-05; First posted 2018-03-21 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Vaccination
MeSH Terms: interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMVAMUNE® (Experimental): Two subcutaneous vaccinations with 0.5 mL IMVAMUNE® vaccine administered at a 4 week intervals
  Interventions: Biological: IMVAMUNE®

INTERVENTIONS:
Biological: IMVAMUNE® — IMVAMUNE® liquid -frozen, containing 1 x 10E8 TCID50 MVA-BN® per 0.5 mL dose

SUMMARY:
Prophylactic smallpox vaccination for personnel actively working with or in the vicinity of replicating vaccinia virus

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18-65 years, who will work with or in the vicinity of a replicating vaccinia virus and who volunteer for the program. Subjects may be vaccinia-naïve or vaccinia-experienced.
* Women of child-bearing potential (WOCBP) must have a negative urine pregnancy test within 48 hours prior to vaccination.
* WOCBP must have used an acceptable method of contraception for at least 30 days prior to the first vaccination and must agree to use an acceptable method of contraception during the vaccination period until at least 28 days after the last vaccination. A woman is considered of child-bearing potential unless post-menopausal or surgically sterilized. (Acceptable contraception methods are restricted to barrier contraceptives which include Food and Drug Administration (FDA)-approved spermicides, intrauterine contraceptive devices, or licensed hormonal products.)
* Read, signed and dated Informed Consent Form.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Uncontrolled serious infection i.e., not responding to antimicrobial therapy.
* History of or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement are not excluded.
* Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; uncontrolled diabetes mellitus; moderate to severe kidney impairment or post organ transplant subjects.
* History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure.
* History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor.
* History of allergies or reactions to eggs, egg products, or gentamycin.
* Having received any vaccinations or planned vaccinations with a live vaccine within 28 days or a killed vaccine within 14 days prior to or after IMVAMUNE®vaccination.
* Chronic administration (defined as more than 6 days) of systemic corticosteroids within 30 days of the first planned vaccination.
* Use of any investigational or non-registered drug or vaccine other than IMVAMUNE® within 30 days preceding the first vaccine dose.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-04-22 (Actual); Primary Completion 2014-11-14 (Actual); Study Completion 2014-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Fujimoto, MD, Principal Investigator — Palo Alto Medical Foundation
Locations (1):
- Palo Alto Medical Foundation, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MVA-BN: Two s.c. vaccinations with 0.5 ml MVA-BN® vaccine containing 1 x 10E8 TCID50 / dose
Period: Overall Study
Arm/Group | MVA-BN
Started | 22
Completed (active trial phase) | 18
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Arm/Group | MVA-BN
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.36 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: ELISA Seropositivity Rate
Description: Seropositivity rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Seropositivity is defined as antibody titers ≥ detection limit (50). Percentages based on number of subjects with data available.
Time Frame: up to Week 7
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MVA-BN
Number analyzed (Participants) | 22
percentage of subjects
  Screening | 40.9 [20.7 to 63.7]
  Week 7 | 100.0 [84.6 to 100.0]

2. Secondary Outcome: ELISA Seroconversion Rate
Description: Seroconversion rate based on Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to the Screening titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: Week 7
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MVA-BN
Number analyzed (Participants) | 22
percentage of subjects | 90.9 [70.8 to 98.9]

3. Secondary Outcome: ELISA GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Titers below the detection limit are included with a value of '1'.
Time Frame: up to Week 7
Population: Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MVA-BN
Number analyzed (Participants) | 22
Titer
  Screening | 370.08 [166.3 to 823.5]
  Week 7 | 14961.54 [11163.8 to 20051.1]

4. Secondary Outcome: Serious Adverse Events
Description: Incidence, relationship and intensity of any Serious Adverse Event (SAE).
Time Frame: up to 32 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN
Number analyzed (Participants) | 22
Participants | 0

5. Secondary Outcome: Related Grade >=3 Adverse Events
Description: Incidence of any Grade >=3 Adverse Events possibly, probably or definitely related to the trial vaccine
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN
Number analyzed (Participants) | 22
Participants | 1

6. Secondary Outcome: Non-serious AEs
Description: Incidence of non-serious AEs
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN
Number analyzed (Participants) | 22
Participants | 19

ADVERSE EVENTS:
Time Frame: up to 32 weeks
Arm/Group | MVA-BN
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 19/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MVA-BN (N=22)
Fatigue (General disorders) | 4
Injection site erythema (General disorders) | 8
Injection site induration (General disorders) | 6
Injection site pain (General disorders) | 15
Injection site pruritis (General disorders) | 4
Injection site swelling (General disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes